CLINICAL TRIAL: NCT05062473
Title: Hypertension Control in the Age of COVID-19: Utilizing Telemedicine for Hypertension Treatment Lifestyle Modification in Central Harlem
Brief Title: Utilizing Telemedicine for Hypertension Treatment Lifestyle Modification in Central Harlem
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-10022836; 1 T1NHP391850100. (Other Grant/Funding Number: Health Resources and Services Administration of the U.S. Department of Health and Human Services)
Record Dates: First submitted 2021-09-02; First posted 2021-09-30 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypertension telemedicine curriculum (Other): All participants participate in the 12-week telemedicine curriculum. All participants will be asked to record their steps via pedometer and their blood pressure measurements via automatic blood pressure arm cuff.
  Interventions: Behavioral: Lifestyle Modification Webinars Focused on Hypertension Control

INTERVENTIONS:
Behavioral: Lifestyle Modification Webinars Focused on Hypertension Control — Participation in a 12-week health education telemedicine curriculum

SUMMARY:
The purpose of this study is to test the feasibility of creating a health education telemedicine curriculum that can be delivered by Weill Cornell Medicine faculty and medical students and NY-Presbyterian Hospital resident physicians to community dwelling adults in an under-resourced local community.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than or equal to 18 years of age.
* Self-report of a hypertension diagnosis.

Exclusion Criteria:

* Pregnant or breastfeeding.
* End-stage renal disease on hemodialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Participant's Satisfaction with the Curriculum at 12 Weeks | Week 12
  Participant's satisfaction with the curriculum will be measured via 5-point Likert scale survey that was created by our research team. Scores will range from a low of "Strongly disagree" to a high of "Strongly agree."
Change in Number of Participants Virtually Attending the Health Education Seminars | Baseline to 12 weeks.
  Virtual attendance to the health education seminars will be collected. The number of participants who virtually attend all health education seminars over the 12 week period will be collected and change in number of participants attending will be assessed.
Change in Participant's Rate of Completion of Weekly Blood Pressure Recordings | Baseline to 12 weeks.
  Participant's rate of completion of the weekly blood pressure recording logs will be measured and analyzed.
Change in Participant's Rate of Completion of Weekly Steps Recordings | Baseline to 12 weeks.
  Participant's rate of completion of the weekly step recording logs will be measured and analyzed.

SECONDARY OUTCOMES:
Mean Change in Systolic Blood Pressure Measurement. | Baseline to week 12
  Participants will self-report weekly up to 4 blood pressure readings taken at baseline through week 12 with their automatic blood pressure arm cuff. The change in systolic blood pressure measurements in this time frame will be assessed.
Mean Change in Diastolic Blood Pressure Measurement. | Baseline to week 12
  Participants will self-report weekly up to 4 blood pressure readings taken at baseline through week 12 with their automatic blood pressure arm cuff. The change in diastolic blood pressure measurements in this time frame will be assessed.
Mean Change in Number of Daily Steps Measured by Pedometer. | Baseline to week 12
  Participants will self-report weekly the number of steps taken as measured by their wrist pedometer at baseline through week 12.
Change in Self-Reported Health Attitudes and Behaviors As Assessed by Survey. | Baseline, week 12
  The name of the survey is " Knowledge, attitudes, and perceptions towards hypertension and cardiovascular disease." The survey was adapted from the Centers for Disease Control and Prevention Behavioral Risk Factor Surveillance System. It consists of both quantitative and qualitative questions assessing participants' demographics, participants' knowledge and attitudes about diet and exercise, and participants' knowledge about hypertension and other related cardiac diseases (i.e. stroke, coronary artery disease). The survey will be administered at enrollment and post-intervention at week 12. Pre- and post-surveys will be compared for accuracy of answers and change in self-reported behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy K Paul, MD, Principal Investigator — Weill Cornell Medicine/NY Presbyterian Hospital
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Artinian NT, Washington OG, Templin TN. Effects of home telemonitoring and community-based monitoring on blood pressure control in urban African Americans: a pilot study. Heart Lung. 2001 May-Jun;30(3):191-9. doi: 10.1067/mhl.2001.112684. PMID 11343005
- [Background] Liu S, Brooks D, Thomas SG, Eysenbach G, Nolan RP. Effectiveness of User- and Expert-Driven Web-based Hypertension Programs: an RCT. Am J Prev Med. 2018 Apr;54(4):576-583. doi: 10.1016/j.amepre.2018.01.009. Epub 2018 Feb 16. PMID 29456025
- [Background] Bove AA, Homko CJ, Santamore WP, Kashem M, Kerper M, Elliott DJ. Managing hypertension in urban underserved subjects using telemedicine--a clinical trial. Am Heart J. 2013 Apr;165(4):615-21. doi: 10.1016/j.ahj.2013.01.004. Epub 2013 Mar 6. PMID 23537980
- See also: Hypertension Hospitalizations and Related Morbidity in New York City — https://www1.nyc.gov/assets/doh/downloads/pdf/epi/databrief83.pdf